CLINICAL TRIAL: NCT06723990
Title: Prospective Observational Monocentric Study to Evaluate the Impact of the HER2DX Assay on Treatment Decisions in Patients With Early Stage HER2+ Breast Cancer: the HER2-BREAST-DX
Brief Title: Evaluation of HER2DX Assay on Treatment Decisions in Patients With Early Stage HER2+ Breast Cancer: the HER2BREASTDX
Acronym: HER2BREASTDX
Status: Recruiting | Type: Observational
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: UID 4259
Record Dates: First submitted 2024-11-27; First posted 2024-12-09 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer Early Stage Breast Cancer (Stage 1-3)
Keywords: HER2 positive breast cancer patients with stage I-III

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NEOADJUVANT SETTING: Neoadjuvant standard treatment for HER2+: A→Tax +T/P
  Interventions: Drug: Neoadjuvant standard treatment for HER2+
- ADJUVANT SETTING: Adjuvant standard treatment for HER2+ (N0): Tax + T (+/-ET); Adjuvant standard treatment for HER2+ (N+): A→Tax +T/P (+/- ET)
  Interventions: Drug: Adjuvant standard treatment for HER2+

INTERVENTIONS:
Drug: Neoadjuvant standard treatment for HER2+ — NEOADJUVANT SETTING
  Groups: NEOADJUVANT SETTING
Drug: Adjuvant standard treatment for HER2+ — ADJUVANT SETTING
  Groups: ADJUVANT SETTING

SUMMARY:
To prospectively evaluate the impact of HER2DX on the decision-making processes of the treating physicians and especially among the routine multidisciplinary tumour board, in defining type and setting of systemic therapy administration in patients with stage I-III HER2+ BC, and the degree of clinician's confidence in the treatment recommendation.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age;
* Histologically confirmed HER2+ breast cancer;
* Stage I-III breast cancer without evidence of distant metastases;
* Being candidate to neoadjuvant/adjuvant therapy and locoregional treatment (surgery +/- radiotherapy);
* Written informed consent, signed by the patient, to study-specific procedures (the consent will consist of 2 levels: level 1 specifically for patients enrolled in the primary endpoint cohort and level 2 for all patients);

Exclusion Criteria:

* HER2- BC;
* Stage IV breast cancer;
* Lack of informed consent because of patient's incapable of discernment or unwilling to participate;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HER2 positive breast cancer patients with stage I-III
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Impact of HER2DX on the decision-making processes of the treating physicians and multidisciplinary tumour board, in patients with stage I-III HER2+ BC | from baseline to the end of treatment at 12 month
  To prospectively evaluate the impact of HER2DX on the decision-making processes of the treating physicians and especially among the routine multidisciplinary tumour board, in defining type and setting of systemic therapy administration in patients with stage I-III HER2+ BC, and the degree of clinician's confidence in the treatment recommendation.

CONTACTS AND LOCATIONS:
Overall Officials: Paola Zagami, Principal Investigator — Istituto Europeo di Oncologia
Locations (1):
- Istituto Europeo di Oncologia, Milan, Italy, Italy